CLINICAL TRIAL: NCT03929146
Title: Randomized Trial Comparing Interscalene Nerve Block to Liposomal Bupivacaine For Pain Management Following Reverse Total Shoulder Arthroplasty (RTSA)
Brief Title: Liposomal Bupivacaine Versus Interscalene Nerve Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Adam Schumaier, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-7698
Record Dates: First submitted 2019-04-15; First posted 2019-04-26 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal Bupivacaine (Experimental): Patients in this group will receive a single intra-operative injection of liposomal bupivacaine near the surgical site (40 ml total: consisting of 20 ml 1.3% liposomal bupivacaine and 20 ml normal saline).
  Interventions: Drug: Exparel
- Interscalene Nerve Block (Other): Patients in this group will receive a single pre-operative interscalene nerve block in the neck/shoulder consisting of 30 ml 0.5% ropivacaine.
  Interventions: Procedure: Interscalene Nerve Block

INTERVENTIONS:
Drug: Exparel — Patients will receive a local injection of liposomal bupivacaine near the end of their shoulder arthroplasty operation.
  Arms: Liposomal Bupivacaine
Procedure: Interscalene Nerve Block — Patients will undergo a pre-operative interscalene nerve block performed by the anesthesiology team.
  Arms: Interscalene Nerve Block

SUMMARY:
The aim of this study is to compare two different pain management interventions in patients undergoing reverse total shoulder arthroplasty. The two interventions are 1) pre-operative interscalene nerve block and 2) intraoperative injection of liposomal bupivacaine (Exparel, Pacira Pharmaceuticals, Parsippany NJ). Specifically, the primary aims of this study are to compare these two interventions on the following: post-operative opioid consumption, pain scores, and patient satisfaction. Additionally, the investigators want to determine if psychological factors, catastrophizing and resilience, are associated with post-operative pain control and satisfaction. The investigators' hypothesis is that the two interventions will have similar pain control efficacy and that the liposomal bupivacaine group will experience faster post-operative recovery, earlier discharge, and improved satisfaction. The investigators also expect patient catastrophizing and resilience to significantly predict the degree of post-operative pain and level of patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* patients who are older than 18 years
* patients undergoing reverse total shoulder arthroplasty

Exclusion Criteria:

* pregnancy
* inability to provide informed consent
* deemed unreliable for follow-up survey completion
* individuals who do not speak English
* those who have an allergy to the study medications (ropivicaine, bupivicaine) or have clinically significant hepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption | 72 hours post-operatively
  Post-operative use of opioid pain medications, measured in morphine equivalents (higher scores are worse)
Visual Analog Scale Pain Scores | 72 hours post-operatively
  Post-operative level of pain measured from 0 (no pain) to 10 (worst pain)
Patient Satisfaction: Rating | 72 hours post-operatively
  Rating of satisfaction with post-operative pain management from 0 (least satisfied) to 10 (most satisfied)
Relationship between catastrophizing, pain, and patient satisfaction | Catastrophizing will be measured pre-operatively
  The effect of patient catastrophizing (measured using the Pain Catastrophizing Scale) on post-operative pain control and satisfaction. The Pain Catastrophizing Scale measures how individuals psychologically respond to pain and hardship, and it ranges from a minimum score of 0 to a maximum score of 52. Higher scores on the Pain Catastrophizing Scale indicate more catastrophic thinking. The patients' catastrophizing scores will be correlated with their post-operative pain scores and their satisfaction scores. A correlation closer to -1 or 1 (correlations range from -1 to 1) indicates a stronger relationship between catastrophizing with pain control and satisfaction.
Relationship between resilience, pain, and patient satisfaction | Resilience will be measured pre-operatively
  The effect of patient resilience (measured using the Brief Resilience Scale) on post-operative pain control and satisfaction. The Brief Resilience Scale measures how individuals psychologically respond to pain and hardship, and it ranges from a minimum score of 1 to a maximum score of 5. Higher scores on the Brief Resilience Scale indicate greater resilience. The patients' resilience scores will be correlated with their post-operative pain scores and their satisfaction scores. A correlation closer to -1 or 1 (correlations range from -1 to 1) indicates a stronger relationship between resilience with pain control and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Schumaier, MD, Principal Investigator — University of Cincinnati, Department of Orthopaedics and Sports Medicine
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No